CLINICAL TRIAL: NCT00720070
Title: A Multi-centre Randomised Phase III Trial Comparing PET-CT Guided Watch and Wait Policy Versus Planned Neck Dissection for the Management of Locally Advanced (N2/N3) Nodal Metastases in Patients With Head and Neck Squamous Cancer
Brief Title: PET/CT Scan-Guided Watchful Waiting or Neck Dissection of Locally Advanced Lymph Node Metastases in Treating Patients Undergoing Chemotherapy and Radiation Therapy for Primary Head And Neck Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Warwick Medical School (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Diagnostic
Other Study IDs: CDR0000597895; WMS-PET-NECK; ISRCTN13735240; EU-20856; MREC-07/Q1604/35; UKCRN ID: 3799
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-12

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage I verrucous carcinoma of the oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage II verrucous carcinoma of the oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage III verrucous carcinoma of the oral cavity; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Magnetic Resonance Spectroscopy

ARMS (2):
- Arm I (Experimental): Patients receive standard concurrent chemoradiotherapy (CRT). Patients undergo PET/CT scan at 9-13 weeks after completion of CRT. Patients with complete response of primary site undergo neck dissection within 4 weeks.
  Interventions: Procedure: positron emission tomography/computed tomography; Procedure: therapeutic conventional surgery
- Arm II (Active Comparator): Patients undergo neck dissection and receive standard concurrent CRT. Patients undergo PET/CT scan at 9-13 weeks after completion of CRT.
  Interventions: Procedure: positron emission tomography/computed tomography; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Procedure: positron emission tomography/computed tomography — Patients undergo PET/CT scan
Procedure: therapeutic conventional surgery — Patients undergo neck dissection

SUMMARY:
RATIONALE: Imaging procedures, such as PET/CT scan, produce pictures of areas inside the body and may help doctors detect residual disease and plan the best treatment. Neck dissection is surgery to remove lymph nodes and other tissues in the neck. It is not yet known whether a neck dissection should always be performed in treating patients with head and neck cancer.

PURPOSE: This randomized phase III trial is studying PET/CT scan-guided watchful waiting compared with neck dissection of locally advanced lymph node metastases in treating patients who are undergoing chemotherapy and radiation therapy for primary head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the efficacy, in terms of overall survival, disease-specific survival, recurrence, quality of life, and cost-effectiveness, of a PET/CT scan-guided watch and wait policy with the current practice of planned neck dissection in the management of advanced (N2 or N3) nodal metastases in patients with primary head and neck squamous cell carcinoma undergoing chemoradiotherapy.
* To assess the predictive value of PET/CT scanning in detecting persistent or residual disease in the primary site.

OUTLINE: This is a multicenter study. Patients are stratified according to center, chemotherapy schedule (concurrent platinum vs concurrent cetuximab vs neoadjuvant and concurrent platinum vs neoadjuvant docetaxel, platinum, and fluorouracil with concurrent platinum), T stage (T1-T2 vs T3-T4), and N stage (N2a-N2b vs N2c-N3). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive standard concurrent chemoradiotherapy (CRT). Patients undergo PET/CT scan at 9-13 weeks after completion of CRT. Patients with complete response of primary site undergo neck dissection within 4 weeks.
* Arm II: Patients undergo neck dissection and then receive standard CRT. Patients undergo PET/CT scan at 9-13 weeks after completion of CRT.

Patients are assessed periodically for quality-of-life. Tissue and blood samples collected periodically are stored for future research.

After completion of study treatment, patients are followed monthly for 1 year and then bimonthly for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed head and neck squamous cell carcinoma (HNSCC), including any of the following subtypes:

  * Oropharyngeal
  * Laryngeal
  * Oral
  * Hypopharyngeal
* No primary nasopharyngeal carcinoma
* Must have clinical and CT/MRI evidence of nodal metastases staged N2 (a, b, or c) or N3

  * No occult nodal metastasis (i.e., large nodal metastasis but no proven primary site on clinical assessment)
  * No N1 nodal metastasis
* Planning to receive curative radical concurrent chemoradiotherapy (approved by study) for primary disease

  * Patients undergoing neoadjuvant chemotherapy followed by concurrent chemoradiotherapy are eligible
* Able to undergo neck dissection surgery
* No current resection for primary tumor planned (e.g., resection of tonsil or base of tongue with flap reconstruction [diagnostic tonsillectomy allowed])
* No distant metastases to chest, liver, bones, or other sites

PATIENT CHARACTERISTICS:

* Not pregnant
* No other cancer diagnosis within the past 5 years except basal cell carcinoma or cervical carcinoma in situ

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior treatment for HNSCC
* No concurrent neoadjuvant chemoradiotherapy without concurrent chemotherapy
* No concurrent adjuvant chemotherapy
* No concurrent chemoradiotherapy for palliative purposes
* No concurrent radiotherapy alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2007-09; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival at 2 years
Health economics using quality adjusted life years

SECONDARY OUTCOMES:
Disease-specific survival
Recurrence and local control in neck
Utility cost
Quality of life
Complication rates
Accuracy of PET-CT scanning for assessing primary tumor

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Mehanna, MD, Principal Investigator — Warwick Medical School
Locations (1):
- Warwick Medical School Clinical Trials Unit, Coventry, England, United Kingdom